CLINICAL TRIAL: NCT06537921
Title: Feasibility Study in Comorbid Obesity and Treatment-Resistant Depression Using Minocycline as Adjunctive Treatment (CODA)
Brief Title: Comorbid Obesity and Depression With an Anti-inflammatory Medication
Acronym: CODA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRAS ID: 333466
Record Dates: First submitted 2024-03-28; First posted 2024-08-05 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Major Depressive Disorder; Inflammation
Keywords: Psychiatry; Immune System; Immunity
MeSH Terms: conditions — Obesity; Depressive Disorder, Major; Inflammation | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: Feasibility
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comorbid depression and obesity (Experimental): Participants with comorbid major depressive disorder (MDD) and obesity (BMI≥30 kg/m2) and c-reactive protein (CRP) levels ≥3mg/L at screening.
  Interventions: Drug: Minocycline 200mg

INTERVENTIONS:
Drug: Minocycline 200mg — Dosage: 2x100mg/daily for 8 weeks

SUMMARY:
Research suggests that only a subset of individuals with major depressive disorder (MDD) may benefit from anti-inflammatory treatments: those who have C-reactive protein (CRP) ≥3 mg/L, a commonly used threshold for "low-grade" inflammation. The emerging link between metabolic and immune abnormalities in MDD suggests that individuals with comorbid obesity and MDD are a subset of people who could particularly benefit from anti-inflammatory treatment. The coexistence of obesity and MDD has been shown to amplify the risk of clinically elevated CRP levels (≥3mg/L). Therefore, people with comorbid obesity, MDD, and CRP ≥3mg/L could be an ideal target population in future randomised clinical trials (RCTs). However, investigation into the feasibility and acceptability of inflammation-targeting treatment in this population is needed first.

Meta-analyses identify minocycline (a tetracycline antibiotic that can cross the blood-brain barrier) as one of the most effective inflammation-targeting medications with antidepressant effects. Minocycline can safely be used long-term at dosages of up to 200mg per day and has low tendency to lead to antibiotic resistance. A pilot RCT of minocycline found a large effect size (Cohen's d=0.98, p<0.001) for the reduction of MDD symptoms compared with placebo. This effect size was even larger (Cohen's d=1.5, p<0.005) in another RCT using minocycline when considering only participants with CRP ≥3mg/L.

One mechanism through which minocycline could ameliorate MDD symptoms appears to involve the activation of indoleamine 2,3-dioxygenase (IDO), which leads to an increase in the expression and function of the serotonin transporter. Studies exploring this anti-inflammatory effect in MDD demonstrate that minocycline indeed can inhibit IDO.

Another pathway through which minocycline could ameliorate MDD symptoms is through the reduction of inflammation at the central level. Minocycline has been shown to reduce microglia activation in preclinical models. Previous literature reports an impact of neuroinflammation on white matter microstructure and brain structure in patients with MDD and in individuals with obesity. Minocycline's effect on white matter structure and myelination has not yet been investigated in humans in vivo. Investigating whether neuroimaging biomarker candidates associated with neuroinflammation could be detected in this study design is needed.

DETAILED DESCRIPTION:
This is a single-centre feasibility using minocycline (200mg/daily) in participants with comorbid obesity and major depressive disorder (MDD). The study aims to investigate the feasibility and acceptability of this proof-of-concept study in comorbid obesity and depression, selected for elevated inflammation, using adjunctive minocycline treatment.

We will test, in a 12-week feasibility, proof-of-concept study, whether individuals with comorbid obesity and treatment-resistant depression will complete an 8-week course of daily minocycline alongside their regular antidepressant treatment, complete biomarker measurements (e.g., blood, saliva, MRI), and complete other outcome measurements (e.g., questionnaires, interviews). Enrolment and retention rates will be monitored over the 12-week period. The acceptability and suitability of all assessment measures will be examined. Participant feedback of their activities will determine the acceptability of this study, and assist refinement of the design in preparation for a future RCT. The study will also aim to provide insight into the feasibility of using biomarkers of inflammation, as well as pathways affected by minocycline, towards the design of a future RCT in individuals with comorbid obesity and depression.

Objective: Determine the feasibility and acceptability of this protocol in comorbid obesity and depression using minocycline as adjunctive treatment.

Minocycline dosing regimen: After successful completion of the Screening Visit (Visit 1), eligible subjects will be invited for the Baseline (Visit 2) when they will be provided with the first bottle of minocycline (oral capsules) lasting 4 weeks. At the 4-week mark, subjects will return to the clinic to complete Visit 3 and associated visit procedures, including returning the medication bottle and any remaining capsules. Upon returning the bottle, the pharmacy will dispense a second bottle for the subject, once again containing minocycline for 4 weeks. In total, subjects will be taking minocycline for 8 weeks. The dose of 200mg will be taken once daily.

Study schedule:

Following consent, participants will be screened to ensure eligibility according to the inclusion and exclusion criteria as well as a small number of assessments (including safety bloods to check liver and kidney functioning) and questionnaires on mood, medical, and psychiatric history. Furthermore, we will ask each participant's general practitioner (GP) for a summary of the participant's medical records (including current and past medications). For females, a pregnancy test will be done at all visits to ensure that they are not pregnant. A small amount of blood (no more than 10ml, or about 2 teaspoons) will be taken to check your levels of inflammation and some other tests to look at overall health and confirm CRP levels are suitably elevated (at least 3mg/L). If following the screening, participants are deemed eligible, they will be invited for a baseline and then Week 4, Week 8, and Week 12 visits. Simultaneously, eligible participants will be sent a saliva sample collection kit in the post to complete at home and bring with them to their next visit. In this kit will be 6 tubes, saliva collection instructions, and a diary to track your sample collections.

At the Baseline (visit 2) visit, we will repeat some of the questionnaires from the previous visit along with some new questionnaires, including some that ask about past stressful events, how they have been feeling since the last visit, and whether any medications have changed. A sample of blood (no more than 50ml, or 3 tablespoons) will be collected to check inflammation levels. At this visit, participants will also undergo their first brain MRI scan lasting approximately an hour. During this visit, participants will be given their first bottle of minocycline by a study doctor. Participants will take 2 capsules (each 100mg) orally, once a day in the mornings with breakfast, for 28 consecutive days, alongside their usual antidepressant. A diary to track the use of minocycline, any side effects or illness, and any medications taken will be provided too, as well as the 2nd saliva sample collection kit to be completed at home.

At Week 4 (visit 3), after 28 days (±3 days) of taking minocycline, participants will return to the clinic for their next assessment. The assessment and blood collection will be the same as those completed at Baseline. No MRI will be conducted here. Participants will also be given their 2nd bottle of minocycline, dose the same as before, to take for another 28 consecutive days. As before, participants should continue taking their antidepressant normally alongside this and continue completing their diary to track the use of minocycline, any side effects, and any other drugs taken. With these, a saliva sample collection kit will again be provided to complete at home.

At Week 8 (visit 4), after another 28 days (±3 days) of taking minocycline, participants will return for their final in-person visit to the clinic. All assessments, including the MRI, will be the same as those conducted at the Baseline visit. The remaining minocycline will be returned to the research team and no new bottle will be dispensed - this is the end of the minocycline administration.

Finally, at Week 12, participants will be contacted by phone to complete the final set of questionnaires - the same set completed in person at the previous visits. No blood or saliva samples will be collected at this time point.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient communication skills to understand the intervention and complete the assessments.
* Able to give informed consent.
* Treatment resistant depressed (i.e., non-responders to current antidepressant treatment, for at least 6-weeks AND at least one other previous antidepressant).
* Tolerant to the current antidepressant.
* Able to undergo 2 MRI scans.
* Accepting augmentation with minocycline.
* CRP >3mg/L at screening.
* No plans to change current therapy for the duration of participation.

Exclusion Criteria:

* Active suicidal ideation.
* Current primary diagnosis of psychotic disorder, bipolar disorder, obsessive-compulsive disorder, or post-traumatic stress disorder.
* Have an acute infection or an autoimmune disorder, because of both the rare but described association between minocycline and systemic lupus erythematosus, and the potential confounder effects of these conditions on immune biomarkers.
* Alcohol misuse disorder or drug addiction.
* Neurological disorders (Parkinson's, Alzheimer's).
* Current serious cardiovascular problems.
* Have acne or psoriasis.
* Currently taking any antibiotic, immunosuppressive medication, or warfarin.
* Taken any tetracycline within the last month.
* Currently taking Lithium or retinoids (Acitretin, Alitretinoin, Isotretinoin).
* Refuse that we contact their GP to inform them about their participation.
* [OPTIONAL - if not met, cannot undergo the MRI] Has any metal implants in their body such as pacemakers, dental fillings, IUD device (if applicable), or had any accidents where metal fragments might have entered the body or eye.
* Pregnant or breastfeeding
* Have a positive pregnancy test before starting the study/are unwilling to take a pregnancy test and are unwilling to agree to use an acceptable form of contraceptive throughout the study period (e.g., condoms, intrauterine device (IUD)/intrauterine system (IUS), injection, patch, ring). Female participants who use combined oral contraceptives as their main form of birth control will need to use an additional barrier method for the duration of treatment and for 7 days following completion of treatment.
* Are currently participating in another Clinical Trial of Investigational Medicinal Product (CTIMP).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Enrolment rate | Throughout recruitment and screening period
  Percentage of participants who consent at the Screening Visit who begin their 8-week course of minocycline.
Intervention adherence | 8 weeks
  Percentage of participants who complete, in full, the 8-week course of minocycline, alongside their usual antidepressant, and the accompanying medication diary. (N=35)
Outcome and Biomarker Measurements | 8 weeks + 12 week follow-up
  Percentage of participants who complete all outcome measurements (i.e., interviews and questionnaires), blood and saliva sample collections (N=35), and all MRI procedures (N=15) at all time points.
Effect size calculations | 12 weeks
  Effect size calculation and power calculation for a range of blood-based and neuroimaging biomarkers changes to inform the design of a future randomised clinical trial (RCT).

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom